CLINICAL TRIAL: NCT01414530
Title: Effects of Oral Contraceptive on Muscle or Joint Ache in Women During Menopausal Transition
Brief Title: Oral Contraceptive During Menopausal Transition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Byung-Koo Yoon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-03-018
Record Dates: First submitted 2011-06-28; First posted 2011-08-11 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Perimenopause
MeSH Terms: interventions — Contraceptives, Oral; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral contraceptive (Experimental)
  Interventions: Drug: oral contraceptive
- NSAID (Active Comparator)
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: oral contraceptive — ethinyl estradiol 0.03mg/levonorgestrel 0.15mg daily for 8 weeks
  Other Names: Minivora
  Arms: oral contraceptive
Drug: NSAID — ibuprofen 200mg/arginine 185mg twice per day for 8 weeks
  Other Names: Carol-F
  Arms: NSAID

SUMMARY:
Muscle or joint pain is one of the most common symptoms during menopausal transition. As this could be severe enough to affect social and daily life and to reduce quality of life, attentions should be paid about this.

Although understanding of muscle or joint pain related to menopause is still insufficient, estrogen can play an important role. Previous studies have shown that estrogen protects cartilage in both animals and humans.

However, perimenopause is different from postmenopause, in the point that estrogen is still secreted with a great fluctuation.

Until now, no study has been performed to evaluate the effects of oral contraceptive on muscle or joint pain in women during menopausal transition. Moreover, since menopausal symptoms vary according to ethnicity and culture, a study in Korean population is necessary.

Therefore, this randomized controlled trial was designed to evaluate the effects of oral contraceptive on muscle or joint pain in women during menopausal transition, compared to NSAID (non-steroidal anti-inflammatory drug).

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women aged 45 or more
* Women who have multiple joint or muscle pain for at least 3 months (at least two sites out of upper and lower extremities or axial)

Exclusion Criteria:

* Rheumatoid arthritis, ankylosing spondylitis, rheumatic polymyalgia, Inflammatory myopathy
* pregnancy
* History of hysterectomy or bilateral oophorectomy
* Vasomotor symptoms
* History of surgery of musculoskeletal system
* History of cancer
* Abnormalities of thyroid function
* Focal neurologic deficit
* Smoking within 1 year
* Uncontrolled hypertension
* Coronary heart disease
* Diabetes mellitus
* Stoke
* Active thromboembolism
* Undiagnosed vaginal bleeding
* Acute hepatic dysfunction
* Gastrointestinal ulcer
* Severe renal dysfunction
* Hypersensitivity to drugs
* Current hormone user or past users within 3 months

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
improvement in symptoms | Eight weeks
  evaluated by fibromyalgia impact questionnaire and visual analogue scale

SECONDARY OUTCOMES:
quality of life | Eight weeks
  evaluated by SF-12

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea